CLINICAL TRIAL: NCT04730050
Title: A Phase I, First-In-Human, Randomized, Double Blind, Placebo Controlled, Single Ascending-Dose and Multi Ascending Dose Study of TT-01025-CL in Healthy Subjects
Brief Title: A Phase I Clinical Trial to Investigate the Safety, Tolerability, and Pharmacokinetic Characteristics of TT-01025-CL in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TT01025US01
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: TT-01025-CL (Experimental): TT-01025-CL
  Interventions: Drug: TT-01025-CL
- Drug: Placebo (Placebo Comparator): Placebo of TT-01025-CL
  Interventions: Drug: TT-01025-CL

INTERVENTIONS:
Drug: TT-01025-CL — Oral tablet

SUMMARY:
To assess the safety, tolerability and pharmacokinetic characteristics of TT-01025 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Age ≥ 18 years and ≤ 55 years, male or female.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, and weighs at least 50 kg.
* No clinically significant findings in medical examination, including physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory tests.
* Male participant and his female spouse/partner who is of childbearing potential agree to use highly effective contraception* consisting of two forms of birth control (at least one of which must be a barrier method) from signing of informed consent throughout the study period and for 90 days after final study drug administration.
* A female subject of childbearing potential who is sexually active agrees to use highly effective contraception* consisting of two forms of birth control (at least one of which must be a barrier method) from signing of informed consent throughout the duration of the study period and for 90 days after last study drug administration. If the next menstrual period is delayed, a pregnancy test will be required for exclusion of pregnancy.

  * Highly effective contraception is defined as:

    * Established use of oral, injected, or implanted hormonal methods of contraception
    * Placement of an intrauterine device or intrauterine system
    * Barrier methods of contraception: condom with spermicidal foam, gel, film, cream, suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, or suppository
* Able to understand and sign informed consent and to comply with the protocol

Exclusion Criteria:

* Any history of clinically serious disease.
* Any active or unstable clinically significant medical condition as judged by the investigator.
* Subject has abnormal Screening findings or Day -2 laboratory value that suggest a clinically significant underlying disease.
* Hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes.
* Received any investigational drug within 30 days or 5x T1/2 whichever is longer before the Screening.
* Participants who have undergone major surgery ≤ 2 months prior to start study drug.
* Impaired cardiac function including clinically significant arrhythmias or clinically significant abnormality in clinical test, including but not limited to any of the following at Screening and

Check-in, repeat testing is allowed for verification, at the discretion of the Investigator:

* Heart rate < 45 beats per minute (bpm) or > 90 bpm (taken during blood pressure measurement).
* Systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg; diastolic blood pressure (DBP) < 50 mmHg or > 90 mmHg.
* Average of the 3 QT intervals corrected using Fridericia's formula (QTcF) > 450 milliseconds.
* Second degree or higher Atrioventricular block on ECG
* Estimated glomerular filtration rate (eGFR) < 90 ml/min/1.73m2

  * Impaired renal function or abnormal liver enzymes at baseline, including but not limited to:
* Alanine aminotransferase (ALT) > upper limit of normal (ULN)
* Aspartate aminotransferase (AST) > ULN
* Estimated glomerular filtration rate (eGFR) < 90 ml/min/1.73m2

  * Women who are pregnant or lactating, or intending to become pregnant before, during or within 90 days after exit from this study.
  * Women with baseline FSH ≥40mIU/ml
  * Participant who has had a loss of more than 100 mL blood (e.g., a blood donation) within 2 months before study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before Check-in, or plans to donate blood, ova or sperm during the study or within 3 months after the study.
  * Participant who has a known history of, or a positive test result for, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) types 1 or 2 at screening.
  * Participant who has used prescription or over-the-counter (OTC) medication (other than ≤2 g/day paracetamol [acetaminophen] or ≤800 mg/day ibuprofen), vitamins, or herbal remedies, within 7 days or 5 half-lives before study drug administration, whichever is longer.
  * Participant who has a history of alcohol abuse (defined as an alcohol intake more than 21 units per week) or a history of drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the investigator. A unit of alcohol is defined as 240 mL of beer, 120 mL of wine, or 20 mL of spirits.
  * Participant who smokes cigarettes or uses other nicotine-containing products (e.g., vape, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers), has done so in the 3 months prior to screening.
  * Consumption of caffeine or xanthine-containing food or beverages from at least 72 hours prior to Check-in to the clinical research unit until at least 24 hours after last drug administration
  * Participant who has a positive test for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, MDMA, oxycodone, phencyclidine, methamphetamine, tricyclic antidepressants, opiates, methadone, cocaine, cannabinoids, amphetamines, or cotinine) at Screening or Check-in.
  * Subject is unable to complete this study for other reasons or the Investigator believes that he or she should be excluded.
  * Participant who has a positive swab test of COVID-19 from Screening or Check-in testing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 30 days

SECONDARY OUTCOMES:
Cmax | up to 7 days post-dose
AUC | up to 7 days post-dose
Terminal half-life | up to 7 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Las Vegas Clinical Research Unit, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No